CLINICAL TRIAL: NCT07175922
Title: Evaluation of csgA Prevalence, Gene Expression and Week-to-Week Variability in Participants With Parkinson's Disease and a History of Gastrointestinal Dysfunction
Brief Title: Research Into the Expression of the csgA-gene and How it Changes in Patients With Parkinson's Disease
Status: Recruiting | Type: Observational
Sponsor: Vertero Therapeutics (Industry)
Responsible Party: Sponsor
Other Study IDs: AXL-5006-001
Record Dates: First submitted 2025-07-22; First posted 2025-09-16 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-09

CONDITIONS: Parkinsons Disease (PD)
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study seeks to understand the prevalence and variability of a gut bacteria gene called csgA in people with Parkinson's Disease. This understanding could inform development of potential new therapies targeting the gut in Parkinson's Disease.

DETAILED DESCRIPTION:
Parkinson's Disease (PD) is a neurodegenerative disorder traditionally associated with motor and non-motor symptoms due to the loss of dopaminergic neurons in the nervous system. Recent research highlights two primary progression patterns: body-first and brain-first PD. In brain-first, PD begins with alpha-synuclein (aSyn) pathology in the brain, particularly in areas like the substantia nigra or olfactory bulb, before potentially involving peripheral systems. Conversely, in the body-first subtype, pathological aSyn aggregates are thought to originate in the enteric nervous system or peripheral autonomic structures, such as the gut and cardiac structures, before spreading to the brain via the vagus nerve. In this subtype of PD, gut dysbiosis and bacterial amyloids could trigger misfolding of aSyn in the enteric nervous system, initiating a cascade of pathology that spreads retrogradely to the brain via the vagus nerve.

The potential influence of the gut microbiome on PD development and progression offers the potential for microbiome targeted therapies to be developed. csgA encodes the major protein subunit of curli, a functional amyloid protein assembly produced by certain gut bacteria like Escherichia coli. Curli proteins help establish extracellular biofilms, and their structural similarity to human amyloids, such as aSyn, suggests they may contribute to pathological processes in PD. csgA protein could therefore be a potential target for therapies. To develop such interventions, understanding the prevalence of csgA within the microbiomes of the PD population and the variability of csgA mRNA expression in individual patients is critical because this information will help determine if csgA mRNA expression can be used to assess a pharmacodynamic effect of a potential therapy. This study therefore focuses on studying the prevalence of csgA in the PD population and the week-to-week intra- and inter-individual variability of csgA mRNA expression.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of PD within 10 years from the time of ICF signing
* A history of gastrointestinal (GI) dysfunction or constipation prior to PD diagnosis at the discretion of the investigator based on screening assessment
* All participants must understand and provide written informed consent prior to any study specific procedures
* Able to speak, read, and understand study procedures in Dutch sufficiently to allow completion of all study assessments

Exclusion Criteria:

* Any known GI disorder if deemed clinically significant by the investigator. GI disorders may include, but are not limited to: Crohn's disease, ulcerative colitis, celiac disease, irritable bowel syndrome, or lactose intolerance
* Recent GI infection in the past 3 months if deemed clinically significant by the investigator.
* Major GI surgery (excluding appendectomy/cholecystectomy), such as bariatric surgery, gastrectomy, esophagectomy, vagotomy, small intestine surgeries, any type of colectomy, colostomy and anorectal surgeries if deemed clinically significant by the investigator

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a diagnosis of Parkinson's disease within the last 10 years in the Netherlands
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-09-25 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
csgA DNA | Baseline stool sample
  Part A: The prevalence of detectable csgA DNA in stool samples from participants diagnosed with Parkinson's disease, as measured by polymerase chain reaction (PCR).
csgA mRNA | Weekly variability assessed over 4 weeks.
  Part B: The intra-individual and inter-individual variability in stool csgA mRNA expression, measured over time, as measured by PCR.

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Human Drug Research, Leiden, Netherlands

IPD SHARING:
Plan to Share IPD: No